CLINICAL TRIAL: NCT02616510
Title: Primary Ovarian Insufficiency, Polycystic Ovary Syndrome & the CardiOvascular Risk Profile
Acronym: POPCORn
Status: Completed | Type: Observational
Sponsor: UMC Utrecht (Other)
Collaborators: Amsterdam UMC, location VUmc (Other); Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Bart CJM Fauser, professor, UMC Utrecht
Other Study IDs: 13-010
Record Dates: First submitted 2015-11-20; First posted 2015-11-30 (Estimated); Last update posted 2018-12-11 (Actual); Status verified 2018-12

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — plasma, serum, urine
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- PCOS: Rotterdam criteria (at least 2 out of three criteria present) oligo-anovulation polycystic ovarian morphology hyperandrogenism
  Interventions: Procedure: cardiovascular screening
- POI: amenorrhea of at least 4 months prior to age 40 years, with follicle stimulating hormone (FSH) levels above 40 IU/L
  Interventions: Procedure: cardiovascular screening

INTERVENTIONS:
Procedure: cardiovascular screening — cardiovascular screening: serum, urine, ECG, carotid intima media thickness (IMT), cardiac ultrasound

SUMMARY:
The polycystic ovary syndrome (PCOS) is the most common endocrinopathy amongst women of reproductive age. PCOS is associated with various cardiovascular risk factors such as obesity, glucose intolerance, dyslipidemia hypertension and the metabolic syndrome. Whether these increased cardiovascular risk factors result in the development of actual cardiovascular disease in later life remains to be established.

Women with premature ovarian insufficiency (POI), experience menopause prior to the age of 40 years. Women with POI may exhibit dyslipidemia. A young age at menopause has been previously associated with increased cardiovascular morbidity and mortality.

DETAILED DESCRIPTION:
Cardiovascular risk profile will be assessed in women with PCOS and POI > 45 years of age, consisting of:

fasting serum and urine analyses blood pressure, length, weight, waist circumference, hip circumference ECG carotid intima media thickness cardiac ultrasound

spare serum, plasma and urine will be stored in -80 degrees celsius biobank.

ELIGIBILITY:
Inclusion Criteria:

* age above 45 years

Exclusion Criteria:

* none

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: women with PCOS according to rotterdam criteria (2 or more of these criteria)
  * oligo/anovulation
  * polycystic ovarian morphology
  * hyperandrogenism
  Women with POI amenorrhea of at least 4 months prior to age 40 years with FSH levels above 40 IU/L
Sampling Method: Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2013-07; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
carotid intima media thickness | 10 years post diagnosis
  ultrasound measurement of thickness of carotid wall (mean IMT), presence of atherosclerotic plaques (yes/no, location)

SECONDARY OUTCOMES:
dyslipidemia | 10 years post diagnosis
  serum measurement of low density lipoprotein cholesterol, triglycerides, total cholesterol, high density lipoprotein cholesterol
insulin and glucose levels | 10 years post diagnosis
C-reactive protein | 10 years post diagnosis
homocysteine | 10 years post diagnosis
uric acid | 10 years post diagnosis
androgen levels | 10 years post diagnosis
electrocardiogram (ECG) | 10 years post diagnosis
  documentation of heart rythm, potential signs of ischemia (ST segment), length PR, QRS, QT, RR interval
cardiac ultrasound (hypertrophy) | 10 years post diagnosis
  measurement of left ventricular ejection fraction and left ventricular mass,

CONTACTS AND LOCATIONS:
Overall Officials: Bart Fauser, prof, Principal Investigator — UMC Utrecht
Locations (1):
- University Medical Center Utrecht, Utrecht, Netherlands

REFERENCES:
- [Derived] Gunning MN, Meun C, van Rijn BB, Daan NMP, Roeters van Lennep JE, Appelman Y, Boersma E, Hofstra L, Fauser CGKM, Rueda-Ochoa OL, Ikram MA, Kavousi M, Lambalk CB, Eijkemans MJC, Laven JSE, Fauser BCJM; CREW consortium. The cardiovascular risk profile of middle age women previously diagnosed with premature ovarian insufficiency: A case-control study. PLoS One. 2020 Mar 5;15(3):e0229576. doi: 10.1371/journal.pone.0229576. eCollection 2020. PMID 32134933
- [Derived] Daan NM, Muka T, Koster MP, Roeters van Lennep JE, Lambalk CB, Laven JS, Fauser CG, Meun C, de Rijke YB, Boersma E, Franco OH, Kavousi M, Fauser BC. Cardiovascular Risk in Women With Premature Ovarian Insufficiency Compared to Premenopausal Women at Middle Age. J Clin Endocrinol Metab. 2016 Sep;101(9):3306-15. doi: 10.1210/jc.2016-1141. Epub 2016 Jun 14. PMID 27300572